CLINICAL TRIAL: NCT01643668
Title: Phase II Study of Reduced Intensity Conditioning With Busulfan/Clofarabine Followed by Allogeneic Stem Cell Transplantation
Brief Title: Busulfan/Clofarabine + Allogeneic Stem Cell Transplantation
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Responsible Party: Principal Investigator, Yi-Bin A. Chen, MD, Principal Investigator, Massachusetts General Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 12-128
Record Dates: First submitted 2012-06-12; First posted 2012-07-18 (Estimated); Results first posted 2017-07-13 (Actual); Last update posted 2017-07-13 (Actual); Status verified 2017-06

CONDITIONS: Acute Myeloid Leukemia; Acute Lymphoblastic Leukemia; Myelodysplastic Syndrome
MeSH Terms: conditions — Leukemia, Myeloid, Acute; Precursor Cell Lymphoblastic Leukemia-Lymphoma; Myelodysplastic Syndromes | interventions — Busulfan; Clofarabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- BuClo RIC + SCT (Experimental): Busulfan and Clofarabine (BuClo) reduced intensity conditioning (RIC) followed by allogeneic stem cell Transplantation (SCT)
  Interventions: Drug: Busulfan; Drug: Clofarabine; Procedure: Allogeneic Stem Cell Infusion

INTERVENTIONS:
Drug: Busulfan — Busulfan as part of reduced intensity conditioning prior to allogeneic stem cell transplantation
Drug: Clofarabine — Clofarabine as part of reduced intensity conditioning prior to allogeneic stem cell transplantation
Procedure: Allogeneic Stem Cell Infusion — Allogeneic stem cell transplantation after reduced intensity conditioning with busulfan / clofarabine chemotherapy

SUMMARY:
This research is a phase II clinical trial. Phase II clinical trials test the effectiveness of an investigational intervention to learn whether it works in treating a specific cancer. "Investigational" means that the study intervention is still being studied and that research doctors are trying to find out more about it. It also means that the FDA has not yet approved this study intervention for your type of cancer.

All participants on this study are treated in an identical manner. The investigators are doing this study because there continues to be a significant risk of relapse of disease after reduced intensity transplantation. In studies which have compared transplants using high-doses of chemotherapy and/or radiation versus reduced intensity transplants, patients undergoing reduced intensity transplants appear to have higher rates of relapse, but lower rates of toxicity and complication. This study attempts to utilize clofarabine, a newer chemotherapy agent shown to be quite active in AML, ALL, and MDS, to increase the anti-tumor effects of the conditioning regimen without accumulating unacceptable toxicity.

The reduced intensity allogeneic stem cell transplantation procedure involves giving you chemotherapy in relatively less intense doses to suppress your immune system. This is followed by an infusion of healthy blood stem cells from a matched related donor or a matched unrelated volunteer donor. It is hoped that these donor cells can eventually then attack any cancer cells which remain.

In this research study, the investigators are looking to see how well this new combination of busulfan and clofarabine works in reduced intensity allogeneic stem cell transplantation. By "works" the investigators mean to analyze safety, ability of donor cells to engraft (take hold), as well as measures of complications including toxicity, infections, graft-vs-host disease (GVHD), and relapse.

DETAILED DESCRIPTION:
You will start the conditioning regimen, which is also called the preparative regimen. Conditioning is done to kill more cancer cells which may remain as well as prepare your body for transplant. You will receive the conditioning drugs into a vein. The conditioning regimen consists of the following drugs: Busulfan and Clofarabine.

While you are in the hospital you will have regular physical exams and you will be asked specific questions about any problems that you might be having. You will also have blood tests every day to look at how your bone marrow is recovering, to give possible transfusional support, and how to see how your liver and kidneys are functioning.

You will receive the following drugs before and after the allogeneic stem cell transplant: Neupogen (G-CSF) injections, drugs to prevent infections, Tacrolimus to prevent GVHD and Methotrexate.

You will have routine and regular follow-up in the transplant clinic after discharge from the hospital. The following will be performed at each visit:

Physical exam to monitor your health and check for signs of GVHD, infections and any side effects you may be having; Blood draw for routine blood tests to measure your blood cell count and chemistry; Blood tests to see if the transplanted stem cells are being accepted and are growing in the body (engraftment); Bone marrow biopsy to see the status of the underlying disease (to be done around 100 days after the stem cell transplant).

You will be asked to return to the clinic, at a minimum, for follow-up visits at 6 months, 9 months, 12 months, 18 months and 24 months after your stem cell transplant.

ELIGIBILITY:
Inclusion Criteria:

* Must have well-matched adult donor willing to donate peripheral blood stem cells with well-matched defined as 8/8 matched related or unrelated donor
* Adequate organ functioning

Exclusion Criteria:

* Pregnant or breastfeeding
* Psychiatric disease severely impairing the compliance of the patient to participate in the study and/or give informed consent
* Evidence of prior exposure to HIV or HCV

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 34 (Actual)
Dates: Start 2012-07; Primary Completion 2016-08 (Actual); Study Completion 2016-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Yi-Bin Chen, MD, Principal Investigator — Massachusetts General Hospital
Locations (3):
- United States (3):
  - Massachusetts General Hospital, Boston, Massachusetts
  - Brigham and Women's Hospital, Boston, Massachusetts
  - Dana-Farber Cancer Institute, Boston, Massachusetts

RESULTS

PARTICIPANT FLOW:
Groups:
- BuClo RIC + SCT: BuClo RIC SCT
  Busulfan: Busulfan as part of reduced intensity conditioning prior to allogeneic stem cell transplantation
  Clofarabine: Clofarabine as part of reduced intensity conditioning prior to allogeneic stem cell transplantation
  Allogeneic Stem Cell Infusion: Allogeneic stem cell transplantation after reduced intensity conditioning with busulfan / clofarabine chemotherapy
Period: Overall Study
Arm/Group | BuClo RIC + SCT
Started | 34
Completed | 33
Not Completed | 1
Not completed — Death | 1

BASELINE CHARACTERISTICS:
Arm/Group | BuClo RIC + SCT
Number analyzed (Participants) | 34
Age, Continuous [Median (Full Range); unit: years] | 63.5 [25 to 74]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9
  Male | 25
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 34
Diagnosis [Count of Participants; unit: Participants]
  Acute Myeloid Leukemia (AML) | 25
  Myelodysplastic Syndrome (MDS) | 5
  Acute Lymphoblastic Leukemia (ALL) | 4
Hematopoietic Cell Transplantation (HCT) Refined Disease Risk Index (DRI) [Count of Participants; unit: Participants] — Categorization of disease risk determined by the Refined Disease Risk Index (DRI) for patients receiving Hematopoietic Cell Transplantation (HCT).
  Participants
    Low | 1
    Intermediate | 27
    High | 6
Disease Stage [Count of Participants; unit: Participants] — Disease stage at time of treatment:
  * CR1: Absence of disease following initial treatment
  * CR2: Complete remission occurs achieved following progression of disease after initial complete remission
  * Partial remission/active disease/ blasts >5%: participants who are not currently in remission
  Participants
    First Complete Remission (CR1) | 25
    Second Complete Remission (CR2) | 6
    Partial remission/active disease/blasts >5% | 3
Cytogenics for patients with AML/MDS [Count of Participants; unit: Participants] — Southwest Oncology Group Risk Stratification Population: The 30 participants diagnosed with ALL or MDS
  Participants
    Favorable: number analyzed (Participants) | 30
    Favorable | 1
    Intermediate: number analyzed (Participants) | 30
    Intermediate | 24
    Adverse: number analyzed (Participants) | 30
    Adverse | 5
ALL Cytogenics [Count of Participants; unit: Participants] — Population: The four participants diagnosed with ALL
  Participants
    Philadelphia Chromosome: number analyzed (Participants) | 4
    Philadelphia Chromosome | 2
    Other: number analyzed (Participants) | 4
    Other | 2
Hematopoietic cell transplantation specific comorbidity index (HCT-CI) [Median (Full Range); unit: units on a scale] — The HTC-CI provides information about the overall and non-relapse mortality risk a patient is likely to experience following a hematopoietic cell transplantation. Lower scores represent lower risk and higher scores represent higher risk. The score is produced by adding up the number of specific risk factors a patient has and can range from 0 to 26. The index is usually characterized as risk categories from 0 to 4+ with patients with four or more risk factors considered high risk.
  units on a scale | 1 [0 to 9]
Donor Type [Count of Participants; unit: Participants] — Matched = Human Leukocyte Antigen (HLA) matched; Related = donor and recipient are genetic relatives
  Participants
    Matched Related | 11
    Matched Unrelated | 23
Cytomegalovirus Serostatus [Count of Participants; unit: Participants]
  Either donor or host positive for virus | 22
  Both negative for virus | 12

OUTCOME MEASURES:

1. Primary Outcome: Assessment of Donor Stem Cell Engraftment: ANC Count
Description: Patients are considered to have achieved donor cell engraftment if they have an absolute neutrophil count (ANC) of at least 500 cells/uL of blood for 3 consecutive measurements and at least 75% of hematopoietic elements are donor-derived as determined by chimerism assays from peripheral blood prior to day +40 after Busulfan/Clofarabine (BuClo) reduced intensity allogeneic stem cell transplantation
Time Frame: 1, 2, 3, and 4 weeks after transplantation
Population: One participant experienced early death before engraftment. Outcome measure was assessed among the remaining 33 evaluable participants.
Measure: Count of Participants; unit: Participants
Groups:
- Treatment Arm: Reduced Intensity Conditioning with Busulfan/Clofarabine followed by Allogeneic Stem Cell Transplantation (BuClo RIC SCT)
  Busulfan: Busulfan as part of reduced intensity conditioning prior to allogeneic stem cell transplantation
  Clofarabine: Clofarabine as part of reduced intensity conditioning prior to allogeneic stem cell transplantation
  Allogeneic Stem Cell Infusion: Allogeneic stem cell transplantation after reduced intensity conditioning with busulfan / clofarabine chemotherapy
Arm/Group | Treatment Arm
Number analyzed (Participants) | 33
Participants
  Neutrophil Engraftment Achieved | 33
  Neutrophil Engraftment Not Achieved | 0

2. Primary Outcome: Donor Stem Cell Engraftment: Platelet Count
Description: Platelet recovery was defined as having a platelet count of at least 20,000 platelets/uL of blood on 2 consecutive measurements without transfusional support prior to day +100 after BuClo RIC HSCT.
Time Frame: 1, 2, 3, 4, 8, and 14 weeks post transplant
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment Arm
Number analyzed (Participants) | 33
Participants
  Platelet Engraftmnet Achieved | 33
  Platelet Engraftmnet Not Achieved | 0

3. Secondary Outcome: Cumulative Incidence of Non-relapse Mortality
Description: The percentage of participants that experienced non-relapse mortality (NRM) at day 100 and 1 year after BuClo RIC SCT. Non-relapse mortality is any mortality that is not associated with or proceeded by disease progression of prior cancers.
Time Frame: 100 days, 1 year
Measure: Number (95% Confidence Interval); unit: percentage of participants who died
Arm/Group | Treatment Arm
Number analyzed (Participants) | 34
percentage of participants who died
  100 Days | 5.9 [1.0 to 17.4]
  1 Year | 24 [13 to 39]

4. Secondary Outcome: Progression-Free and Overall Survival
Description: The 1-year and 2-year progression-free and overall survival measured from the time of stem cell transplantation. Progression is the recurrence or increase in the number of cancer cells found in the body.
Time Frame: 1 year, 2 years
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Treatment Arm
Number analyzed (Participants) | 34
percentage of participants
  Progression Free Survival at 1 year | 50 [32 to 65]
  Progression Free Survival at 2 years | 50 [32 to 65]
  Overall Survival at 1 year | 56 [38 to 71]
  Overall Survival at 2 years | 56 [38 to 71]

5. Secondary Outcome: Cumulative Incidence and Severity of Acute GVHD Within 100 Days Post Transplant
Description: The percentage of participants who experienced grades 2-4 and grades 3-4 acute graft-versus-host disease (GVHD) by 100 days post transplantation. GVHD is a condition that can occur following an allogenic stem cell transplantation when the donated bone marrow or peripheral stem cells view the recipients body as foreign and the donated cell/marrow attack the body. Acute GVHD is generally observed within the first 100 days post transplant. Acute GVHD is associated with increased treatment related morbidity and mortality. Grade I GVHD is characterized as mild disease, grade II GVHD as moderate, grade III as severe, and grade IV life-threatening. The grade of the GVHD is determined by grading GHVD associated adverse events. Associated adverse events were graded using Common Terminology Criteria for Adverse Events (CTCAE) version 4 which uses the same mild, moderate, severe, life threatening grading system as the overall GHVD assessment.
Time Frame: 100 days
Measure: Number (95% Confidence Interval); unit: percentage of Participants
Arm/Group | Treatment Arm
Number analyzed (Participants) | 34
percentage of Participants
  Grades II-IV acute GVHD | 21 [8.9 to 35.6]
  Grades III-IV acute GVHD | 12 [3.6 to 25.1]

6. Secondary Outcome: Cumulative Incidence of Chronic GVHD at One Year
Description: The percentage of participants who experienced chronic Graft Versus Host Disease (GVHD) by one year. GVHD is a condition that can occur following an allogenic stem cell transplantation when the donated bone marrow or peripheral stem cells view the recipients body as foreign and the donated cell/marrow attack the body. Chronic GVHD normally occurs after the first 100 days post transplantation. Chronic GVHD can adversely influence long term survival.
Time Frame: 1 year
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Treatment Arm
Number analyzed (Participants) | 34
percentage of participants | 44 [27 to 60]

7. Secondary Outcome: Incidence of Hepatic Veno-occlusive Disease
Description: The number of participants that experienced hepatic veno-occlusive disease (VOD). VOD is a condition in which some of the small veins in the liver are obstructed.
Time Frame: 2 years
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment Arm
Number analyzed (Participants) | 34
Participants | 0

8. Secondary Outcome: Grade 3 or 4 Toxicities
Description: The number of participants that experienced the specified grade 3 and 4 non-hematological toxicities during treatment and follow-up as assessed by Common Terminology Criteria for Adverse Events version 4(CTAE v 4.0). Grade 3 toxicity is considered to be severe and grade 4 is considered to be life threatening.
Time Frame: 2 years
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment Arm
Number analyzed (Participants) | 34
Participants
  Bacterial Infection | 10
  Viral Infection | 1
  Fungal Infection | 2
  Mucositis | 1
  Increased bilirubin | 1
  Increased alanine aminotransferase | 1
  Increased aspartate aminotransferase | 1
  Engraftment Syndrome | 0
  Febrile Neutropenia | 2
  Sepsis | 1
  Acute Renal Failure | 1
  Diffuse alveolar hemorrhage | 0
  Idiopathic pneumonia syndrome | 0

9. Secondary Outcome: Infection-related Complications
Description: The number of patients with infection-related complications
Time Frame: 2 years
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment Arm
Number analyzed (Participants) | 34
Participants | 0

ADVERSE EVENTS:
Time Frame: Duration of the study, median duration of 20 months
Description: Adverse events were assessed from the start of reduced intensity conditioning with Busulfan/Clofarabine until the participant died, relapsed/ had progressive disease, was taken off the study, or withdrew consent (median duration of 20 months). Adverse events were assessed at every study visit. Adverse events were assessed with the use of physicals/review of systems and routine laboratory tests.
Arm/Group | Treatment Arm
All-Cause Mortality (participants affected / at risk) | 15/34
Serious Adverse Events (participants affected / at risk) | 14/34
Other Adverse Events (participants affected / at risk) | 24/34
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment Arm (N=34)
Acute Kidney Injury (Renal and urinary disorders) | 1 (1)
Alanine aminotransferase increased (Investigations) | 1 (1)
Anemia (Blood and lymphatic system disorders) | 1 (1)
Blood bilirubin increased (Investigations) | 1 (1)
Erythroderma (Skin and subcutaneous tissue disorders) | 1 (1)
Hypertension (Vascular disorders) | 1 (1)
Hypertriglyceridemia (Metabolism and nutrition disorders) | 1 (1)
Lung Infection (Infections and infestations) | 1 (1)
Neutrophil Count Decreased (Investigations) | 3 (3)
Platelet count decreased (Investigations) | 1 (1)
Respiratory Failure (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Sepsis (Infections and infestations) | 1 (1)
Viral Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment Arm (N=34)
Abdominal pain (Gastrointestinal disorders) | 1 (1)
Activated partial thromboplastin time prolonged (Investigations) | 1 (1)
Acute kidney injury (Renal and urinary disorders) | 1 (1)
Alanine aminotransferase increased (Investigations) | 1 (1)
Anal mucositis (Gastrointestinal disorders) | 1 (1)
Anemia (Blood and lymphatic system disorders) | 4 (7)
Anorexia (Metabolism and nutrition disorders) | 2 (2)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1)
Aspartate aminotransferase increased (Investigations) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 2 (2)
Blood bilirubin increased (Investigations) | 3 (3)
Depression (Psychiatric disorders) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 1 (1)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Erythroderma (Skin and subcutaneous tissue disorders) | 1 (1)
Fatigue (General disorders) | 1 (2)
Febrile neutropenia (Blood and lymphatic system disorders) | 2 (2)
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 4 (5)
Glucose intolerance (Metabolism and nutrition disorders) | 1 (1)
Hemoglobin increased (Investigations) | 1 (1)
Hip fracture (Injury, poisoning and procedural complications) | 2 (2)
Hyperglycemia (Metabolism and nutrition disorders) | 1 (1)
Hypertension (Vascular disorders) | 3 (3)
Hyponatremia (Metabolism and nutrition disorders) | 1 (1)
Lung infection (Infections and infestations) | 3 (3)
Mucositis oral (Gastrointestinal disorders) | 1 (1)
Muscle weakness lower limb (Musculoskeletal and connective tissue disorders) | 1 (1)
Myalgia (Musculoskeletal and connective tissue disorders) | 1 (1)
Nausea (Gastrointestinal disorders) | 3 (3)
Neoplasms benign, malignant and unspecified (incl cysts and polyps) - Other, specify (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Neutrophil count decreased (Investigations) | 5 (5)
Palmar-plantar erythrodysesthesia syndrome (Skin and subcutaneous tissue disorders) | 1 (2)
Platelet count decreased (Investigations) | 4 (5)
Renal and urinary disorders - Other, specify (Renal and urinary disorders) | 1 (1)
Skin infection (Infections and infestations) | 1 (1)
Thromboembolic event (Vascular disorders) | 1 (1)
Weight loss (Investigations) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes